CLINICAL TRIAL: NCT04800627
Title: A Phase I/II Trial of Pevonedistat in Combination With Pembrolizumab in Patients With dMMR/MSI-H Cancers
Brief Title: Pevonedistat and Pembrolizumab for the Treatment of dMMR/MSI-H Metastatic or Locally Advanced Unresectable Solid Tumor
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per PI
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1065; NCI-2020-13862 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1065 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-01-12; First posted 2021-03-16 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pembrolizumab; pevonedistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pevonedistat, pembrolizumab) (Experimental): Patients receive pevonedistat IV over 60 minutes on days 1, 3, and 5, and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Pevonedistat

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Pevonedistat — Given IV
  Other Names: MLN4924; Nedd8-Activating Enzyme Inhibitor MLN4924

SUMMARY:
This phase I/II trial identifies the side effects and best dose of pevonedistat when given together with pembrolizumab in treating mismatch repair deficiency (dMMR)/high-frequency microsatellite instability (MSI-H) solid tumor that has spread to other places in the body (metastatic) or has spread to nearby tissue or lymph nodes (locally advanced) and cannot removed by surgery (unresectable). Pevonedistat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving pevonedistat and pembrolizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine safety and phase II dose of pevonedistat in combination with pembrolizumab. (Phase I) II. To assess the efficacy of pevonedistat in combination with pembrolizumab in patients with dMMR/MSI-H cancers.

SECONDARY OBJECTIVES:

I. To assess additional efficacy endpoints of the combination of pevonedistat and pembrolizumab in dMMR/MSI-H cancers.

II. To assess the safety of pevonedistat and pembrolizumab in the dMMR/MSI-H patient cohort.

III. To assess the pharmacodynamics impact of pevonedistat and pembrolizumab on tumor and immune-related components.

EXPLORATORY OBJECTIVES:

I. Immune context evaluation of tumor microenvironment. II. Determine clinical benefit. III. Evaluate pevonedistat pharmacokinetics and resistance mechanisms in combination therapy.

OUTLINE: This is a phase I, dose escalation study of pevonedistat followed by a phase II study.

Patients receive pevonedistat intravenously (IV) over 60 minutes on days 1, 3, and 5, and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Patients must have metastatic or locally advanced unresectable solid tumor
* Tumor that is deficient in mismatch repair (dMMR) or microsatellite instability high (MSI-H) as determined by one of three methods:

  * Immunohistochemistry determined dMMR by complete loss of MLH1, PMS2, MSH2 or MSH6
  * Polymerase chain reaction (PCR) determined microsatellite instability at > 30% of tested microsatellites
  * Next-generation determined MSI-H based upon instability at multiple microsatellites as determined by the specific next generation sequencing panel
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Hemoglobin >= 8 g/dL (may transfuse to achieve this threshold)
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Albumin > 2.7 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) except in patients with Gilbert's syndrome. Patients with Gilbert's syndrome may enroll if direct bilirubin =< 3 x ULN of the direct bilirubin
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3.0 x ULN
* Creatinine clearance >= 30 mL/min according to MD Anderson standard, automated laboratory calculation
* Human immunodeficiency virus (HIV) patients may be considered as long as they meet the following criteria:

  * CD4 count > 350 cells/mm^3
  * Undetectable viral load
  * No history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR If they are of childbearing potential:
  * Agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug (female and male condoms should not be used together), or
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug (female and male condoms should not be used together), or
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Demonstrated prior progression on or after anti-PD1/L1 based therapy by radiographic progression. The potential for psuedoprogression should be excluded by concurrent tumor marker (for example carcinoembryonic antigen) or circulating tumor deoxyribonucleic acid [ctDNA] elevation, or clinical symptom progression, or short interval repeat imaging confirming progression. (if uncertain if patient meets eligibility please discuss with study principal investigator [PI])

  * Must have received at least 2 doses of a PD1/PD-L1 inhibitor
  * Progressive disease either during therapy or within 2 months of last dose of therapy
* Measurable disease by immune modified Response Evaluation Criteria in Solid Tumors (iRECIST) version (v)1.1 by treating investigator or study PI
* Tumor that is accessible to biopsy and patient is willing to undergone mandatory tumor biopsies at pre-treatment and on-treatment (unless exception granted by study PI)
* Life expectancy >= 12 weeks as judged by treating physician

Exclusion Criteria:

* Treatment with any investigational products within 4 weeks before the first dose of any study drug
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study procedures
* Active uncontrolled infection or severe infectious disease, such as severe pneumonia, meningitis, or septicemia
* Major surgery within 14 days before the first dose of any study drug or a scheduled surgery during study period
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Life-threatening illness unrelated to cancer
* Patients with uncontrolled coagulopathy or bleeding disorder
* Known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection

  * Note: Patients who have isolated positive hepatitis B core antibody (i.e., in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load
* Known hepatic cirrhosis or severe pre-existing hepatic impairment
* Known cardiopulmonary disease defined as:

  * Unstable angina;
  * Congestive heart failure (New York Heart Association [NYHA] Class III or IV);
  * Myocardial infarction (MI) within 6 months prior to first dose (patients who had ischemic heart disease such as a (ACS), MI, and/or revascularization greater than 6 months before screening and who are without cardiac symptoms may enroll);
  * Symptomatic cardiomyopathy;
  * Clinically significant arrhythmia:

    * History of polymorphic ventricular fibrillation or torsade de pointes,
    * Permanent atrial fibrillation [a fib], defined as continuous a fib for >= 6 months,
    * Persistent a fib, defined as sustained a fib lasting > 7 days and/or requiring cardioversion in the 4 weeks before screening,
    * Grade 3 a fib, within 6 months of starting protocol therapy, defined as symptomatic and incompletely controlled medically, and
    * Patients with paroxysmal a fib or < Gr 3 a fib for period of at least 6 months are permitted to enroll provided that their rate is controlled on a stable regimen.
  * Clinically significant pulmonary hypertension requiring pharmacologic therapy
* Uncontrolled high blood pressure (i.e., systolic blood pressure >= 160 mm Hg, diastolic blood pressure >= 100 mm Hg)
* Prolonged rate corrected QT (QTc) interval >= 500 msec, calculated according to institutional guidelines
* Left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiogram or radionuclide angiography
* Known moderate to severe chronic obstructive pulmonary disease, interstitial lung disease, and pulmonary fibrosis
* Known central nervous system (CNS) involvement unless controlled with surgery or radiation therapy and has demonstrated no progression over 3 months from last local modality therapy
* Systemic antineoplastic therapy or radiotherapy for other malignant conditions within 14 days before the first dose of any study drug
* Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on day 1 before first dose of study drug
* Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s)
* Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s)
* Known hypersensitivity to a study agent(s)
* Residual adverse events from prior therapy (other than endocrinopathies or alopecia or neuropathy due to chemotherapy) that have not resolved to grade 0-1
* Serious adverse immune related adverse events (grade 3 or 4) with previous immune checkpoint therapy, that were symptomatic and required prolong immunosuppression (> 6 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Overman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Company stopped development of the drug and shut down the entire program with pevonedistat. Takeda had a negative phase III of the agent in liquid tumors and thus shut the program. It was not due to any toxicity, but lack of path for FDA indication.
Period: Overall Study
Arm/Group | Treatment (Pevonedistat, Pembrolizumab)
Started | 2
Completed | 0
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pevonedistat, Pembrolizumab)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose of Pevonedistat When Combined With Pembrolizumab (Phase I)
Time Frame: 21 days
Population: No data collected due to early termination of the protocol.
Arm/Group | Treatment (Pevonedistat, Pembrolizumab)
Number analyzed (Participants) | 0

2. Primary Outcome: Objective Response (Partial Response [PR] or Complete Response [CR]) (Phase II)
Description: Will be assessed by immune modified Response Evaluation Criteria in Solid Tumors (iRECIST) version (v) 1.1.
Time Frame: Through study completion, an average of 1 year
Population: No data collected due to early termination of the protocol.
Arm/Group | Treatment (Pevonedistat, Pembrolizumab)
Number analyzed (Participants) | 0

3. Secondary Outcome: Changes in Protein Misfolding
Description: Will analyze the pharmacodynamics impact of pevonedistat by evaluating changes in protein misfolding between pre-treatment and on-treatment tumor biopsies.
Time Frame: Up to 24 weeks
Population: No data collected due to early termination of the protocol.
Arm/Group | Treatment (Pevonedistat, Pembrolizumab)
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Will be assessed by iRECIST v1.1. Will be estimated using the method of Kaplan and Meier.
Time Frame: Through study completion, an average of 1 year
Population: No data collected due to early termination of the protocol.
Arm/Group | Treatment (Pevonedistat, Pembrolizumab)
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Response
Time Frame: Through study completion, an average of 1 year
Population: No data collected due to early termination of the protocol.
Arm/Group | Treatment (Pevonedistat, Pembrolizumab)
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival
Description: Will be estimated using the method of Kaplan and Meier.
Time Frame: Through study completion, an average of 1 year
Population: No data collected due to early termination of the protocol.
Arm/Group | Treatment (Pevonedistat, Pembrolizumab)
Number analyzed (Participants) | 0

7. Secondary Outcome: Incidence of Adverse Events
Time Frame: Through study completion, an average of 1 year
Population: No data collected due to early termination of the protocol.
Arm/Group | Treatment (Pevonedistat, Pembrolizumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after the last dose of study medication up to 1 year
Arm/Group | Treatment (Pevonedistat, Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Company stopped development of the drug and shut down the entire program with pevonedistat. Takeda had a negative phase III of the agent in liquid tumors and thus shut the program. It was not due to any toxicity, but lack of path for FDA indication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT04800627/Prot_SAP_000.pdf